CLINICAL TRIAL: NCT04816136
Title: Consequences of Post Stroke Polysomnographic Abnormalities on Functionnal Recovery and Survival After an Ischemic Stroke
Acronym: PSG-AVC
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0120
Record Dates: First submitted 2021-03-19; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Ischemic Stroke; Cerebral Infarct; Sleep Apnea; Periodic Limb Movement Disorder
Keywords: Functional recovery; Ischemic stroke / cerebral infarct; Sleep; Polysomnography
MeSH Terms: conditions — Ischemic Stroke; Cerebral Infarction; Sleep Apnea Syndromes; Nocturnal Myoclonus Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with a sleep recording performed: patients with a sleep recording performed in the sleep unit in Montpellier University Hospital, who had an ischemic stroke before the recording.
  Interventions: Other: Sleep recording (already done)

INTERVENTIONS:
Other: Sleep recording (already done) — Sleep recording (already done)

SUMMARY:
Ischemic stroke is a major public health issue, likely to cause functional disability. It is well known that sleep has an impact on brain plasticity, and after an ischemic stroke, studies have shown subjective sleep quality alterations and sleep architecture abnormalities.

Furthermore, there is no clear guideline showing the usefulness of a systematic sleep investigation following an ischemic stroke.

The aim of the study is to identify retrospectively correlation between polysomnographic abnormalities (sleep apnea, periodic limb movements, disturbed sleep architecture…) and functional recovery after an ischemic stroke. The study also assesses the impact of sleep abnormalities on survival, and the risk of new cardiovascular event.

DETAILED DESCRIPTION:
This study is a retrospective observational study, from a cohort of patients who had a sleep recording (polysomnography or ventilatory polygraphy performed in Montpellier University Hospital) following an ischemic stroke.

ELIGIBILITY:
Inclusion criteria:

* men and women, more than 18 years old
* medical history of ischemic stroke
* who had a sleep recording following the stroke

Exclusion criteria:

* others types of strokes (bleeding, transient ischemic attack, cerebal veinous thrombosis)
* patients less than 18 years old

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients selected with computer codes of disease and examination corresponding to the criteria : sleep recording and ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Correlation between polysomnographic abnormalities and functional recovery | functional recovery at 6 months
  polysomnographic abnormalities : sleep apnea, periodic limb movements, distribution of sleep stage / functional recovery : modified rankin score and National Institutes of Health Stroke Scale at 6 months

SECONDARY OUTCOMES:
Correlation between polysomnographic abnormalities and survival, onset of new cardio vascular events, functionnal recovery and quality of life. | survival or onset of new cardio vascular events at one year, quality of life evaluated by self questionnaire at one year and functionnal recovery (modified rankin score and National Institutes of Health Stroke Scale) at one year
  polysomnographic abnormalities : sleep apnea, periodic limb movements, distribution of sleep stage / survival or onset of cardio vascular events, quality of life (SF 36), modified rankin score and National Institutes of Health Stroke Scale at one year.

CONTACTS AND LOCATIONS:
Overall Officials: Yves DAUVILLIERS, MD PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC